CLINICAL TRIAL: NCT02239575
Title: Collection of Retrospective (Archival) Samples and Prospective Collection of Surplus Tissue and Blood Samples
Acronym: GBCPRT0009
Status: Withdrawn | Type: Observational
Sponsor: Global BioClinical (Industry)
Responsible Party: Sponsor
Other Study IDs: GBC PRT0009
Record Dates: First submitted 2014-07-16; First posted 2014-09-15 (Estimated); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Cancer
Keywords: Assorted cancers (oncology)
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — pre-surgical blood samples and/or surplus surgical oncology tissues
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will enroll specimens from subjects diagnosed with various cancers and who have either:

1. RETROSPEFCTIVE / ARCHIVAL SAMPLES already undergone surgical resection of their tumor and have one or more formalin fixed and paraffin embedded (FFPE) blocks on file within the local (or affiliated) pathology archive (replicate blocks from same tumor) or blocks no longer required to be maintained on file - discard blocks, or
2. PROSPECTIVE SAMPLES are scheduled to undergo surgical treatment and who prior to scheduled surgery, provide informed consent and donate a 10-20 ml blood sample. After surgery, surplus tissues (including tumor and adjacent normal tissues) not required for diagnosis will be collected.

Subject clinical information will be collected, including basic demographic information, medical history, current cancer history and treatment. A final pathology report will be obtained for each subject's surgical specimen. In some instances, and based on the cancer indications required, longitudinal data may also be collected at a frequency of every 6 months to once per year. Longitudinal data will include information on study subject survival and disease recurrence.

DETAILED DESCRIPTION:
CANCER INDICATIONS:

Bladder Cancer - Urothelial carcinoma - nonpapillary Bladder Cancer - Urothelial carcinoma - papillary Brain Cancer - Astrocytoma Brain Cancer - Glioblastoma Brain Cancer - Medulloblastoma Breast Cancer - Ductal Carcinoma Breast Cancer - Lobular Carcinoma Cervical Cancer - Squamous Cell Carcinoma Colorectal Cancer - Adenocarcinoma Esophageal Cancer - Adenocarcinoma Gastric Cancer Head and Neck Cancer - Squamous Cell Carcinoma Hematologic Cancer - Acute Lymphocytic Leukemia (ALL) Hematologic Cancer - Acute Myeloid Leukemia (AML) Hematologic Cancer - Chronic Lymphocytic Leukemia (CLL) Hematologic Cancer - Diffuse Large B-cell Lymphoma Hematologic Cancer - Multiple Myeloma (MM) Hematologic Cancer - Non-Hodgkins Lymphoma (NHL) Kidney Cancer - Papillary Carcinoma Kidney Cancer - Renal cell Carcinoma Liver Cancer - Hepatocellular Carcinoma Lung Cancer - Adenocarcinoma Lung Cancer - Squamous Cell Cancer Melanoma Pancreatic Cancer - Ductal Adenocarcinoma Prostate Cancer - Adenocarcinoma Sarcomas Thyroid Cancer - Follicular Carcinoma Thyroid Cancer - Papillary Carcinoma Uterine Cancer - Endometrial Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Any adult age
* Any sex
* Able to provide consent for surplus tissue and/or blood donation
* Diagnosed with one of the cancer indications listed below:
* Scheduled to undergo surgical resection of tumor (exception for hematological cancers)
* Have not yet received treatment for cancer

Exclusion Criteria:

* Not diagnosed with required cancer indication
* Not scheduled to undergo surgical resection of the tumor
* Have already received cancer treatment (such as chemotherapy, radiation, surgery) for the current cancer or a previously diagnosed cancer
* Not able to donate an adequate volume of blood to meet minimum requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surplus surgical specimens from subjects diagnosed with cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Identification and validation of cancer biomarkers in archival formalin fixed and paraffin embedded tumor samples | Sample Collection May 2014 to Dec 2016, disease recurrence follow-up periods for upto 1 year
  This study will identify novel cancer biomarkers associated with various solid tumor sub-types, tumor stages, and from patients with various responses to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Mucci, Study Director — GBC
Locations (1):
- Global BioClinical, Seattle, Washington, United States